CLINICAL TRIAL: NCT00132795
Title: Therapeutic IVR to Augment CBT in Alcohol Dependence
Brief Title: Using Telephone Technology to Prevent Relapse After Alcoholism Treatment
Acronym: ATIVR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, John E. Helzer, MD, Professor of Psychiatry, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIAAAHEL014270; R01AA014270 (NIH)
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Alcoholism
Keywords: Cognitive Therapy; Recurrence; Prevention; Educational Technology
MeSH Terms: conditions — Alcoholism; Recurrence | interventions — Ethanol; Secondary Prevention; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Therapeutic Phone System (Experimental): patients assigned to this condition will have unlimited access to the therapeutic telephone system for 4 months.
  Interventions: Behavioral: Daily monitoring of alcohol & drug use, & therapy skills
- 2 Standard care (Active Comparator): Standard post-CBT care (i.e., no formal relapse prevention or professional treatment).
  Interventions: Behavioral: control group

INTERVENTIONS:
Behavioral: Daily monitoring of alcohol & drug use, & therapy skills — Comparison(s): patients completing group CBT for substance abuse will be randomly assigned to two conditions. In one condition, patients will have unlimited access to the therapeutic telephone system for 4 months. The other condition is standard care (i.e., no formal relapse prevention).
  Other Names: relapse prevention
  Arms: 1 Therapeutic Phone System
Behavioral: control group — standard care (no added treatment)
  Arms: 2 Standard care

SUMMARY:
The purpose of this study is to determine whether a telephone based self-help program will prevent relapse among individuals undergoing standard substance abuse treatment.

DETAILED DESCRIPTION:
Relapse rates in the first few months following substance abuse treatment are as high as 50%, in spite of the immediate effectiveness of treatments such as Cognitive Behavioral Therapy (CBT). Continuing use of therapy skills following treatment is associated with maintenance of treatment gains. We have programmed a telephone to deliver pre-recorded summaries and rehearsal sessions of skills learned in therapy. The system also includes monthly feedback messages from therapists. We expect that this ad-lib access to therapy skills would allow patients to generalize skills to their personal post-treatment lives. It would also allow individuals in remote or rural areas to obtain access to assistance without travel barriers.

Comparison(s): patients completing group CBT for substance abuse will be randomly assigned to two conditions. In one condition, patients will have unlimited access to the therapeutic telephone system for 4 months. The other condition is standard care (i.e., no formal relapse prevention).

ELIGIBILITY:
Inclusion Criteria:

* Meets current DSM-IV criteria for alcohol dependence
* Active drinking during the three months prior to entry into treatment
* Minimum age of 19
* Minimum sixth grade reading level.

Exclusion Criteria:

* Meets criteria for a current psychotic illness
* Imminent plans to move or be incarcerated
* Presence of such severe hearing, visual, or cognitive deficit(s) that participation in CBT or use of an Interactive Voice Response (IVR) system are not possible
* Inability to identify at least one "locator" person to assist in tracking for follow-up assessments
* Does not have telephone service within the home
* Incarceration while in active protocol in the study
* Attendance of less than 8 of 12 CBT sessions

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2005-05; Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Amount of alcohol and use | 4 months and one year
  drinks per day, drinks per drinking day, percent days abstinent, heavy drinking days

SECONDARY OUTCOMES:
Utilization of the telephone system components during the study | 4 months and one year
  call rate, access of coping skills reviews and practices, access of monthly messages.

CONTACTS AND LOCATIONS:
Overall Officials: John E. Helzer, MD, Principal Investigator — University of Vermont
Locations (1):
- UVM Health Behavior Research Center, Burlington, Vermont, United States

REFERENCES:
- See also: Investigator's home page — http://www.med.uvm.edu/hbrc/